CLINICAL TRIAL: NCT05931809
Title: Evaluation of the Perception of Quality of Care of Patients Admitted to a Medical-Surgical ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, ICU Assistent Physician, Hospital Sao Domingos
Other Study IDs: HSD 2023 2
Record Dates: First submitted 2023-06-17; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Critically Ill
Keywords: Critically ill patients; Servqual tool; Quality of care; Expectations; Perceptions
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Serqual tool — The SERVQUAL scale will be applied with the questionnaire of expectations in the first 24 hours after admission and perception questionnaire within the first 24 hours after discharge.

SUMMARY:
The objective of this prospective observational cohort study is to describe the perception of quality of care of patients or reference companions admitted to a medical-surgical ICU.

DETAILED DESCRIPTION:
Background: Quality assessment in health systems is essential for the improvement and development of services. Assessments using the structure, process and outcomes model are the most widespread, however understanding the health system as a business model makes assessment essential. how much the service is able to meet the expectations of the patient and the market.

The Institute for Healthcare Improvement (IHI) highlights three domains (Triple aim) in which health systems must develop. Among them is "Improving the patient experience". One of the 6 domains of quality of care is patient-centeredness. Several funding institutions and scientific authorities have, in recent years, encouraged patient-centered clinical research with the use of outcomes that are also patient-centered.

The perception of the quality of the service provided to the critically ill patient or even is an uncommon outcome in the literature, especially evaluated with an objective and effective tool.

The SERVQUAL tool proposed by Parasuraman et al. It aims to compare the expectations and perceptions of the patient/companion regarding the quality of care provided.

In the literature, data on patient-centered perspectives and demands are scarce.

Purpose: To identify the difference between expectation and perception of care quality during the stay in the general ICU of a tertiary hospital. Objectives: To evaluate the perception of quality of care of patients admitted to a general ICU through the SERVQUAL tool translated and culturally adapted to the portuguese idiom.

Methods: A prospective, observational cohort study involving adult patients admitted to the general ICU (53 beds) of a tertiary hospital from July 1 to September 30, 2023. The SERVQUAL tool questionnaire of expectations will be applied in the first 24 hours after admission to the ICU and the perception questionnaire applied in the first 24 hours after discharge from the unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* consent form signed by the patient or a family member.

Exclusion Criteria:

* Patients unable to respond and who do not have reference companions
* Patients readmitted to the ICU during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the 53 beds general ICU during the study period. The SERVQUAL scale will be applied with the questionnaire of expectations in the first 24 hours of admission and perception questionnaire within the first 24 hours after discharge.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Servqual tool | 30 days
  The questionnaire consists of 5 domains with 22 questions graded from 1 to 7 according to perceived quality and expected in each sphere of care delivery. Domains are:
  1. Tangibles. Equipment, physical structure, presentation of professionals and materials.
  2. Reliability. Ability to resolve problems and resolve them within the deadline, and record without errors.
  3. Availability and responsiveness. Ability to inform about the therapeutic plan, to execute on time, availability of professionals to help clients and degree of occupation of professionals to meet demands.
  4. Security / Trust. Ability to inspire security, education of professionals and knowledge of processes by professionals.
  5. Empathy. To provide individual attention, standard opening hours, sincere interest in resolving demands and ability to meet demands individually.
  The result is analyzed with the calculation: Average result of reality - Average result of expectation = Gap of perception of quality of care.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burstin H, Leatherman S, Goldmann D. The evolution of healthcare quality measurement in the United States. J Intern Med. 2016 Feb;279(2):154-9. doi: 10.1111/joim.12471. PMID 26785953
- [Result] Sixma HJ, Kerssens JJ, Campen CV, Peters L. Quality of care from the patients' perspective: from theoretical concept to a new measuring instrument. Health Expect. 1998 Nov;1(2):82-95. doi: 10.1046/j.1369-6513.1998.00004.x. PMID 11281863
- [Result] Jonkisz A, Karniej P, Krasowska D. The Servqual Method as an Assessment Tool of the Quality of Medical Services in Selected Asian Countries. Int J Environ Res Public Health. 2022 Jun 26;19(13):7831. doi: 10.3390/ijerph19137831. PMID 35805492
- [Result] Malathi A, Jasim KM. Validating the relationship between service quality, patient sensitivity and experience towards medical applications using SERVQUAL. Int J Med Inform. 2022 Dec;168:104883. doi: 10.1016/j.ijmedinf.2022.104883. Epub 2022 Oct 5. PMID 36209699
- [Result] Regaira Martinez E, Sola Iriarte M, Goni Viguria R, Del Barrio Linares M, Margall Coscojuela MA, Asiain Erro MC. [Care quality in intensive care evaluated by the patients using a service quality scale (SERVQUAL)]. Enferm Intensiva. 2010 Jan-Mar;21(1):3-10. doi: 10.1016/j.enfi.2009.10.001. Epub 2010 Feb 1. Spanish. PMID 20170830
- [Result] Lu SJ, Kao HO, Chang BL, Gong SI, Liu SM, Ku SC, Jerng JS. Identification of quality gaps in healthcare services using the SERVQUAL instrument and importance-performance analysis in medical intensive care: a prospective study at a medical center in Taiwan. BMC Health Serv Res. 2020 Sep 29;20(1):908. doi: 10.1186/s12913-020-05764-8. PMID 32993641
- [Result] Fan LH, Gao L, Liu X, Zhao SH, Mu HT, Li Z, Shi L, Wang LL, Jia XL, Ha M, Lou FG. Patients' perceptions of service quality in China: An investigation using the SERVQUAL model. PLoS One. 2017 Dec 22;12(12):e0190123. doi: 10.1371/journal.pone.0190123. eCollection 2017. PMID 29272312